CLINICAL TRIAL: NCT02347657
Title: A Phase 3, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous for the F508del CFTR Mutation
Brief Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VX-661 in Combination With Ivacaftor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX14-661-106
Expanded Access: Available
Record Dates: First submitted 2015-01-12; First posted 2015-01-27 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis
Keywords: Homozygous for the F508del CFTR Mutation
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to VX-661 plus IVA FDC tablet administered orally in the morning and placebo matched to IVA tablet administered orally in the evening up to Week 24.
  Interventions: Drug: VX-661 Plus Ivacaftor Combination Placebo; Drug: Ivacaftor placebo
- VX-661/IVA (Experimental): VX-661 100 mg plus IVA 150 mg FDC tablet administered orally in the morning and IVA 150 mg tablet administered orally in the evening up to Week 24.
  Interventions: Drug: VX-661 Plus Ivacaftor Combination; Drug: Ivacaftor

INTERVENTIONS:
Drug: VX-661 Plus Ivacaftor Combination — FDC tablet, oral use
  Arms: VX-661/IVA
Drug: Ivacaftor — Tablet, oral use
  Arms: VX-661/IVA
Drug: VX-661 Plus Ivacaftor Combination Placebo — FDC tablet, oral use
  Arms: Placebo
Drug: Ivacaftor placebo — Tablet, oral use
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double blind, placebo controlled, parallel group, multicenter study in people with cystic fibrosis (CF) who are homozygous for the F508del CF transmembrane conductance regulator (CFTR) gene mutation.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter study in people with CF who are homozygous for the F508del-CFTR mutation. This study is designed to evaluate the efficacy and safety of VX-661 in combination with Ivacaftor (IVA, VX-770). The active treatment regimen comprised of a morning dose of a fixed-dose combination (FDC) tablet of 100 milligram (mg) VX-661/150 mg IVA once daily (qd) and an evening dose of IVA 150 mg to be taken approximately 12 hours after the morning dose. The placebo regimen was visually matched tablets to be taken with the same schedule as the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for the F508del CFTR mutation, genotype to be confirmed at the Screening Visit
* Confirmed diagnosis of CF defined as a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis
* Forced expiratory volume at one second (FEV1) ≥40% and ≤90% of predicted normal for age, sex, and height during screening
* Stable CF disease as judged by the investigator
* Willing to remain on a stable CF medication regimen through Week 24 or, if applicable, the Safety Follow up Visit

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1 (first dose of study drug)
* Pregnant or nursing females (females of childbearing potential must have a negative pregnancy test at Screening and Day 1)
* Sexually active participants of reproductive potential who are not willing to follow the contraception requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (27):
  - Little Rock, Arkansas
  - Long Beach, California
  - Denver, Colorado
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Manchester, New Hampshire
  - Long Branch, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - Rochester, New York
  - Syracuse, New York
  - Akron, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Fort Worth, Texas
  - Tyler, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
- Copenhagen O, Denmark
- France (6):
  - Marseille, Bouches-du-Rhone
  - Roscoff, Finistere
  - Bordeaux, Girande
  - Lille, Nord
  - Paris, Paris
  - Pierre-Bénite, Rhone
- Germany (7):
  - Heidelberg, Baden-Wurttemberg
  - Munich, Bavaria
  - Würzburg, Bavaria
  - Frankfurt am Main, Hesse
  - Giessen, Hesse
  - Belfast, State of Berlin
  - Berlin
- Ireland (2):
  - Cork
  - Dublin
- Italy (5):
  - Genova
  - Palermo
  - Roma
  - Torino
  - Verona
- Netherlands (5):
  - Groningen
  - Nijmegen
  - Rotterdam
  - The Hague
  - Utrecht
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (7):
  - Exeter, Devon
  - Liverpool, Lancashire
  - Sheffield, South Yorkshire
  - Newcastle upon Tyne, Tyne & Wear
  - Birmingham, West Midlands
  - Belfast
  - London

REFERENCES:
- [Derived] Acaster S, Mukuria C, Rowen D, Brazier JE, Wainwright CE, Quon BS, Duckers J, Quittner AL, Lou Y, Sosnay PR, McGarry LJ. Development of the Cystic Fibrosis Questionnaire-Revised-8 Dimensions: Estimating Utilities From the Cystic Fibrosis Questionnaire-Revised. Value Health. 2023 Apr;26(4):567-578. doi: 10.1016/j.jval.2022.12.002. Epub 2022 Dec 9. PMID 36509366
- [Derived] Taylor-Cousar JL, Munck A, McKone EF, van der Ent CK, Moeller A, Simard C, Wang LT, Ingenito EP, McKee C, Lu Y, Lekstrom-Himes J, Elborn JS. Tezacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del. N Engl J Med. 2017 Nov 23;377(21):2013-2023. doi: 10.1056/NEJMoa1709846. Epub 2017 Nov 3. PMID 29099344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 91 sites in 12 countries.
Pre-assignment Details: A total of 510 participants were randomized and 509 participants were treated in the study.
Groups:
- Placebo: Placebo matched to VX-661 plus Ivacaftor (IVA, VX-770) fixed dose combination (FDC) tablet administered orally in the morning and placebo matched to IVA tablet administered orally in the evening up to Week 24.
- VX-661/IVA: VX-661 100 milligram (mg) plus IVA 150 mg FDC tablet administered orally in the morning and IVA 150 mg tablet administered orally in the evening up to Week 24.
Period: Overall Study
Arm/Group | Placebo | VX-661/IVA
Started | 259 | 251
Treated | 258 | 251
Completed | 241 | 236
Not Completed | 18 | 15
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 8 | 4
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Randomized but not treated | 1 | 0
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who carried the intended cystic fibrosis transmembrane conductance regulator (CFTR) allele mutation and had received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-661/IVA | Total
Number analyzed (Participants) | 256 | 248 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (9.5) | 26.9 (11.2) | 26.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 121 | 246
  Male | 131 | 127 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 250 | 234 | 484
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 254 | 245 | 499
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline (Day 1) in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Through Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Day 1, Through Week 24
Population: FAS included all randomized participants who carry the intended CFTR allele mutation and have received at least 1 dose of study drug. Here 'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FEV1
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 256 | 245
Percentage of predicted FEV1 | -0.6 [-1.3 to 0.0] | 3.4 [2.7 to 4.0]
Statistical Analysis 1: Comparison: Placebo vs VX-661/IVA; Testing was performed according to the hierarchical testing procedure to control the overall type I error for tested at α = 0.05; Test type: Superiority; p < 0.0001, Mixed model for repeated measures (MMRM); Least Squares (LS) Mean Difference = 4.0, 95% CI 2-sided [3.1 to 4.8]

2. Secondary Outcome: Relative Change From Baseline (Day 1) in ppFEV1 Through Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Day 1, Through Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 256 | 245
percent change | -0.5 [-1.7 to 0.6] | 6.3 [5.1 to 7.4]
Statistical Analysis 1: Comparison: Placebo vs VX-661/IVA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, MMRM; LS mean difference = 6.8, 95% CI 2-sided [5.3 to 8.3]

3. Secondary Outcome: Number of Pulmonary Exacerbations Per Year
Description: Pulmonary exacerbation was defined as a new event or change in antibiotic therapy for greater than or equal to 4 sinopulmonary signs/symptoms. Pulmonary exacerbation events per year (48 weeks) were reported.
Time Frame: Day 1 through Week 24
Population: FAS included all randomized participants who carry the intended CFTR allele mutation and have received at least 1 dose of study drug.
Measure: Number; unit: pulmonary exacerbation events per year
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 256 | 248
pulmonary exacerbation events per year | 0.99 | 0.64
Statistical Analysis 1: Comparison: Placebo vs VX-661/IVA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0054, Negative Binomial Regression; Event Rate Ratio = 0.65, 95% CI 2-sided [0.48 to 0.88]

4. Secondary Outcome: Absolute Change From Baseline (Day 1) Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilograms (kg) divided by height in square meter (m^2).
Time Frame: Day 1, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram per square meter (kg/m^2)
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 245 | 237
kilogram per square meter (kg/m^2) | 0.12 [0.03 to 0.22] | 0.18 [0.08 to 0.28]
Statistical Analysis 1: Comparison: Placebo vs VX-661/IVA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4127, MMRM; LS mean difference = 0.06, 95% CI 2-sided [-0.08 to 0.19]

5. Secondary Outcome: Absolute Change From Baseline (Day 1) in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 24
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Day 1, Through Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 256 | 246
units on a scale | -0.1 [-1.6 to 1.4] | 5.0 [3.5 to 6.5]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, inpatient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AE that increased in severity or newly developed at or after initial dosing of study drug to Week 28 was considered treatment-emergent.
Time Frame: Day 1 up to Week 28
Population: Safety Set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 258 | 251
Participants
  Participants with AEs | 245 | 227
  Participants with SAEs | 47 | 31

7. Secondary Outcome: Number of Participants With at Least One Pulmonary Exacerbation Pulmonary Exacerbation Through Week 24
Description: Pulmonary exacerbation was defined as a new event or change in antibiotic therapy for greater than or equal to 4 sinopulmonary signs/symptoms. Time to event data was not collected and instead, Number of Subjects with first event were collected and are reported. Time-to-first pulmonary exacerbation was planned to be estimated using Kaplan-Meier (KM) estimates. However, due to less than 50% of events, time-to-first event data was not estimated. Instead, number of participants with at least one pulmonary exacerbation event were collected and are reported.
Time Frame: Day 1 through Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 256 | 248
Participants | 88 | 62

8. Secondary Outcome: Absolute Change From Baseline (Day 1) in Sweat Chloride Through Week 24
Description: Sweat samples were collected using an approved collection device.
Time Frame: Day 1, Through Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 242 | 240
millimole per liter (mmol/L) | 0.2 [-0.8 to 1.2] | -9.9 [-10.9 to -8.9]

9. Secondary Outcome: Absolute Change From Baseline (Day 1) in BMI Z-score at Week 24 in Participants Less Than (<) 20 Years Old at the Time of Screening)
Description: BMI was defined as weight in kg divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score (BMI z-score).
Time Frame: Day 1, Week 24
Population: Analysis population included all randomized participants who received at least 1 dose of study drug and were <20 years of age at the time of screening. Here 'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 74 | 76
z-score | -0.02 [-0.10 to 0.06] | -0.06 [-0.14 to 0.02]

10. Secondary Outcome: Absolute Change From Baseline (Day 1) in Body Weight at Week 24
Time Frame: Day 1, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | VX-661/IVA
Number analyzed (Participants) | 245 | 237
kg | 0.6 [0.3 to 0.9] | 0.7 [0.4 to 1.0]

11. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of VX-661, VX-661 Metabolites (M1 VX-661 and M2-VX-661), Ivacaftor (IVA) and IVA Metabolite (M1-IVA)
Description: This outcome was not planned to be assessed in Placebo arm.
Time Frame: Pre-morning dose on Week 16
Population: Pharmacokinetic (PK) set included all randomized participants who received any amount of study drug and had a PK assessment. Here 'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-661/IVA
Number analyzed (Participants) | 233
nanogram per milliliter (ng/mL)
  VX-661 | 1890 (1150)
  M1 VX-661 | 4730 (1730)
  M2 VX-661 | 4830 (2750)
  IVA | 815 (572)
  M1 IVA | 1590 (961)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Description: Safety Set included all participants who received at least 1 dose of the study drug.
Arm/Group | Placebo | VX-661/IVA
All-Cause Mortality (participants affected / at risk) | 0/258 | 0/251
Serious Adverse Events (participants affected / at risk) | 47/258 | 31/251
Other Adverse Events (participants affected / at risk) | 243/258 | 227/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=258) | VX-661/IVA (N=251)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 32 | 23
Pneumonia (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood glucose abnormal (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=258) | VX-661/IVA (N=251)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 75 | 57
Nasopharyngitis (Infections and infestations) | 39 | 42
Rhinitis (Infections and infestations) | 14 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 83 | 66
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 42 | 36
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 33 | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Abdominal pain (Gastrointestinal disorders) | 22 | 23
Nausea (Gastrointestinal disorders) | 18 | 23
Diarrhoea (Gastrointestinal disorders) | 23 | 17
Vomiting (Gastrointestinal disorders) | 15 | 13
Abdominal pain upper (Gastrointestinal disorders) | 17 | 10
Constipation (Gastrointestinal disorders) | 14 | 7
Pyrexia (General disorders) | 32 | 28
Fatigue (General disorders) | 30 | 16
Headache (Nervous system disorders) | 36 | 44
Alanine aminotransferase increased (Investigations) | 13 | 8
Bacterial test positive (Investigations) | 16 | 8
Rash (Skin and subcutaneous tissue disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT02347657/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02347657/SAP_001.pdf